CLINICAL TRIAL: NCT05155696
Title: A Randomised Controlled Trial of the Effects of a Probiotic Drink on Behaviour, Sleep and the Microbiome in Children With ADHD
Brief Title: Probiotic Supplementation in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's University, Twickenham (Other)
Collaborators: Goldsmiths, University of London (Other); London South Bank University (Other)
Responsible Party: Principal Investigator, Kate, Senior Lecturer in Psychology, St. Mary's University, Twickenham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMU_ETHICS_2020-21_240
Record Dates: First submitted 2021-11-11; First posted 2021-12-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: ADHD
Keywords: microbiome; ADHD; probiotic; Kefir
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomised double-blind quantitative repeated measures design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a randomly generated 6-digit participant code will be allocated to each participant as a unique identifier for all data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kefir probiotic drink (Experimental): Daily kefir for 6 weeks.
  Interventions: Dietary Supplement: Experimental: Kefir probiotic drink (supplied by Nourish)
- placebo comparator (Placebo Comparator): Daily non-fermented dairy based equivalent drink for 6 weeks.
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Experimental: Kefir probiotic drink (supplied by Nourish) — 125ml per day of dairy based probiotic drink (Kefir) containing ≥ 50billion colony forming units (CFU), supplied in plain packaging.
  Arms: Kefir probiotic drink
Dietary Supplement: Placebo comparator — 125ml of non-fermented dairy based placebo (UHT milk) per day, supplied in plain packaging.
  Arms: placebo comparator

SUMMARY:
This randomised, placebo controlled trial explores the effects of supplementation with a probiotic drink (kefir) in children diagnosed with ADHD on behaviour, sleep, attention and the gut microbiome.

DETAILED DESCRIPTION:
Children with Attention Deficit Hyperactivity Disorder (ADHD) can suffer debilitating symptoms, including problematic behaviour and sleep. Dietary manipulations may be a helpful treatment option for children, but the most effective are highly restrictive, with little known about why they might work.

Optimising gut bacteria may help alleviate some of the symptoms of this condition via the gut-brain-axis. The consumption of a probiotic fermented drink (kefir) can positively influence composition of gut bacteria.

The purpose of this study is to explore the effects of supplementation of a probiotic drink (kefir) on behaviour, sleep, attention and the gut microbiome in children diagnosed with ADHD.

In a six-week randomised controlled double-blind, placebo controlled trial, 70 children diagnosed with ADHD (aged 8-13 years) will be randomised to be given either a probiotic drink (kefir) or a placebo drink. At the beginning and the end of the study a combination of questionnaires, cognitive assessment, sleep/physical activity measures and microbiome analysis will be employed to assess the effect of kefir consumption on symptoms of ADHD and the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* A previous diagnosis of ADHD according to the DSM-IV or DSM-V criteria by a qualified health care professional.
* Children aged between 8 and 13 years at the time of study.
* Children with a comorbidity will be accepted.
* Both males and females

Exclusion Criteria:

* Children currently undergoing a current course of behavioural therapy.
* Children with a reported milk allergy or lactose intolerance.
* Reported use of antibiotics, probiotics, antifungals or steroids in the past four weeks.
* Diagnosis of a gastrointestinal disorder e.g., Inflammatory Bowel Disease or Coeliac disease.
* Diagnosis of an auto-immune disease or compromised immunity.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Change in The Strengths and Weakness of ADHD-symptoms and Normal-behaviour (SWAN) scale | week 0 and week 6
  18 item scale comparing the child to other children of the same age. Each item is responded to on a seven-point scale ranging from far below average (-3) to far above average (+3).
  The scores are summed and divided by the number of items, to express the summary score as the average rating-per-item (range -3 to +3, with lower scores indicating more severe ADHD symptoms).

SECONDARY OUTCOMES:
Change in The Go/NoGo test | week 0 and week 6
  Participants respond to a particular stimulus while various stimuli are presented on a computer screen. There are 1500 milliseconds between each response, with 320 repetitions.
  Go errors (errors of omission) - A higher score = greater inattention (worse)
  NoGo errors (errors of commission) - A higher score = greater impulsivity (worse)
  Go reaction times - A higher score = less impulsivity (better)
  Go reaction time variability - A higher score = greater inattention (worse)
Change in mean activity during sleep. | week 0 and week 6
  Actigraphy recordings. Range 0-∞. A higher score = less sound sleep (worse).
Change in minutes spent awake during the down period | week 0 and week 6
  Actigraphy recordings. Range 0-∞. A higher score = less sound sleep (worse).
Change in sleep latency | week 0 and week 6
  Actigraphy recordings of time taken to fall asleep. Range 0-∞. A higher score = more time taken to fall asleep (worse).
Change in sleep efficiency | week 0 and week 6
  Actigraphy recordings of % down period spent asleep, after removing sleep latency. A higher score = better.
Change in wake after sleep onset | week 0 and week 6
  Actigraphy recordings of minutes spent awake during the down period after removing sleep latency. Range 0-∞. A higher score = less sound sleep (worse).
Change in sleep fragmentation | week 0 and week 6
  Actigraphy recordings of the number of awakenings/ total minutes of sleep x 100) - Higher score = more fragmented sleep (worse).
Change in mean daytime activity | week 0 and week 6
  Actigraphy recording of mean daytime activity. (0-∞) not necessarily worse or better.
The Consensus Sleep diary | week 0 and week 6
  Record of sleep - used qualitatively to detect and remove artefacts from the data. Takes approximately 3 minutes per day to complete.
The Consensus Sleep diary | week 6
  Record of sleep - used qualitatively to detect and remove artefacts from the data. Takes approximately 3 minutes per day to complete.
Change in The Child's Sleep habits questionnaire | week 0 and week 6
  Consists of 33 items. Each item is rated by parents using a three-point scale (with some items reverse-scored):
  3 - Usually =occurs 5+ times a week 2 - Sometimes = occurs 2-4 times a week
  1 - Rarely = occurs 0-1 times a week
  A Total Sleep Disturbances score is calculated as the sum of all scored questions.
  Total scores range from 33 to 99 - higher scores indicate more problematic sleep.
Change in Sleep self report | week 0 and week 6
  Consists of 26 items. Each item is rated by children using a three-point scale (with some items reverse-scored):
  3 - Usually = occurs 5+ times a week 2 - Sometimes = occurs 2-4 times a week
  1 - Rarely = occurs 0-1 times a week.
  A Total Sleep Disturbances score is calculated as the sum of all scored questions.
  Total scores range from 26 to 78 - higher scores indicate more problematic sleep.
Change in The Gastrointestinal Severity Index | week 0 and week 6
  A three-point rating scale across six gastrointestinal symptoms. A higher scores indicate worse symptoms.
  Total scores range from 0-12 - higher scores indicating more severe symptoms.
Change in stool microbiome analysis | week 0 and week 6
  Investigate if there are changes in diversity and species in week 6 relative to week 0.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lawrence, PhD, Principal Investigator — St. Mary's University, Twickenham
Locations (1):
- St Mary's University, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
anonymised data will be made available on an open access repository.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and Statistical analysis plan available as soon as protocol is published - no end date to availability.
Access Criteria: Open Access

REFERENCES:
- [Derived] Lawrence K, Fibert P, Toribio-Mateas M, Gregory AM, Hobbs J, Quadt F, Wright S, Cotter PD, Patel S, Myrissa K. Effects of kefir on symptoms, sleep, and gut microbiota in children with ADHD: a randomised controlled trial. BMC Psychiatry. 2025 Nov 24;25(1):1117. doi: 10.1186/s12888-025-07568-8. PMID 41286799
- [Derived] Lawrence K, Fibert P, Hobbs J, Myrissa K, Toribio-Mateas MA, Quadt F, Cotter PD, Gregory AM. Randomised controlled trial of the effects of kefir on behaviour, sleep and the microbiome in children with ADHD: a study protocol. BMJ Open. 2023 Dec 7;13(12):e071063. doi: 10.1136/bmjopen-2022-071063. PMID 38149413